CLINICAL TRIAL: NCT04429633
Title: Strain-based vs. Left Ventricular Ejection Fraction-based Cardiotoxicity Prevention Strategy in Patients With Breast Cancer Who Treated With Adjuvant Trastuzumab
Brief Title: Strain vs. Left Ventricular Ejection Fraction-based Cardiotoxicity Prevention in Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yeon Hee Park, Professor, MD, PhD, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-11-128
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Cardiotoxicity; Breast Cancer; Prevention; Adjuvant; Trastuzumab
MeSH Terms: conditions — Cardiotoxicity; Breast Neoplasms | interventions — candesartan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Cardiac intervention (Active Comparator): Starting candesartan in patients with left ventricular ejection fraction (LVEF) between 45% and 50% by echocardiogram.
  Interventions: Drug: Candesartan
- Early Cardiac intervention (Active Comparator): Starting candesartan in patients with decreased myocardial strain below 18% regardless of LVEF by echocardiogram.
  Interventions: Drug: Candesartan

INTERVENTIONS:
Drug: Candesartan — If GLS decreased less than 18% or LVEF decreased to 45-50% during the treatment of adjuvant trastuzumab, start candesartan medication.

SUMMARY:
Comparing preventive effect of myocardial global longitudinal strain-based cardioprotective stragety (angiotensin receptor blocker prophylaxis) with left ventricular ejection fraction-based strategy in breast cancer patients treated with adjuvant trastuzumab.

DETAILED DESCRIPTION:
Despite the left ventricular global longitudinal strain (GLS) enables early prediction of trastuzumab-related cardiomyopathy, its clinical application has been hampered due to the lack of appropriate evaluation and treatment strategies. Therefore, we aimed to evaluate the effect of early intervention strategy (GLS-based cardiotoxicity monitoring and administration of candesartan) by comparing with conventional intervention strategy (left ventricular ejection fraction-based cardiotoxicity monitoring and administration of candesartan) in breast cancer patients who treated with adjuvant trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Female aged ≥ 18 years
* Pathologically confirmed HER2-positive breast cancer
* Adjuvant treatment plan comprises at least 12 cycles of Trastuzumab
* Baseline echocardiogram should be performed before starting trastuzumab
* Cumulative anthracycline dose ≤ 300mg/m2
* Written informed consent to participate in the study

Exclusion Criteria:

* History of hypersensitivity or alllergic reaction to the study medication
* Metastatic breast cancer
* Treatment with angiotensin converting enzyme(ACE) inhibitor , Angiotensin receptor blocker (ARB), beta-blocking agents, or diuretics
* Patients with NCI/CTCAE grade ≥ 2 congestive heart failure, myocardial infarction, symptomatic left ventricular systolic dysfunction, heart's valve disease (≥ moderate), arrhythmias (Grade ≥ 3) < 12 months before enrollment
* Pregnancy or breast feeding
* Baseline systolic pressure < 90mmHg
* Cumulative anthracycline dose > 300mg/m2
* Serious concurrent illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2019-07-19 (Actual); Primary Completion 2022-07-18 (Estimated); Study Completion 2023-07-18 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (LVEF) | at months 3,6,9,12,18
  Maximum change in LVEF

SECONDARY OUTCOMES:
Overt chemotherapy induced cardiotoxicity | any time
  LVEF < 45%, decline in LVEF by >10% to a value to 45-49%, symptomatic congestive heart failure
Changes in cardiac biomarker | at months 3,6,9,12,18
  NT-pro BNP, cardiac troponin

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea